CLINICAL TRIAL: NCT02632136
Title: Laparoscopic-assisted Transversus Abdominis Plane (TAP) Block for Laparoscopic Total Extra Peritoneal (TEP) Inguinal Hernia Repair: a Prospective, Double-blinded, Randomized, Clinical Trial
Brief Title: Lap TAP Block for Laparoscopic TEP Inguinal Hernia Repair: a Prospective, Double-blinded, Randomized, Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mayo General Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Asif Khan, Registrar, General Surgery, Mayo General Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MGHIreland
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Laparoscopic TAP Block in TEP Inguinal Hernia Repair.
Keywords: Laparoscopic; TAP Block; Total extra peritoneal Inguinal hernia repair
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP block group (Active Comparator): This group will receive 30 ml of 0.25% Bupivacine given as Transversus Abdominus Plane Block under direct Laparascopic view. The TAP block will be injected in the angle of Petit above the anterior superior iliac supine.
  They will also receive normal saline injections at port sites, which will be injected before the ports are inserted. 15 ml of normal saline will be divided in aliquots of 7, 4 and 4 ml. 7 ml will be injected at sub-umblical port side and 4 ml each at the site of other two ports.
  Interventions: Drug: TAP Block Group
- Peri-Portal block Group (Placebo Comparator): They will receive 0.5% Bupivacaine injections at port sites, which will be injected before the ports are inserted. 15 ml of 0.5% Bupivacaine will be divided in aliquots of 7, 4 and 4 ml. 7 ml will be injected at sub-umblical port side and 4 ml each at the site of other two ports.
  This group will also receive 30 ml of Normal Saline Injection given as Transversus Abdominus Plane Block under direct Laparascopic view. The TAP block will be injected in the angle of Petit above the anterior superior iliac supine.
  Interventions: Drug: Peri-Portal Block Group

INTERVENTIONS:
Drug: TAP Block Group — Transversus Abdominus Plane (TAP) block: Bupivacaine (30 ml of 0.25%)is injected between internal oblique and transveralis facia. The location of needle and the bleb that is formed after the injection is inspected under diect laparoscopic vision.
  Other Names: 0.25% Bupivacaine
  Arms: TAP block group
Drug: Peri-Portal Block Group — 15 ml of 0.5% Bupivacaine is injected in the skin and subcutaneous tissue before inserting the ports. 7 ml out of it is injected at sub-umblical port and 4 ml each a the site of other two ports.
  Other Names: 0.5% Bupivacaine
  Arms: Peri-Portal block Group

SUMMARY:
A newly developed technique of TAP block solely performed by surgeons will be used for postoperative pain relief following laparoscopic total extra peritoneal (TEP) Inguinal hernia repair. Our alternative hypothesis is that laparoscopic-assisted TAP block is better than the periportal wound infiltration in controlling the postoperative pain.

DETAILED DESCRIPTION:
Hypothesis:

A newly developed technique of TAP block solely performed by surgeons will be used for postoperative pain relief following laparoscopic total extra peritoneal (TEP) Inguinal hernia repair. Our alternative hypothesis is that laparoscopic-assisted TAP block is better than the periportal wound infiltration in controlling the postoperative pain.

Significance of the study:

Postoperative pain control is very important in day case surgery. Use of local anaesthetics has a significant role in this scenario.

No study to date examines the use of laparoscopically delivered TAP blocks in TEP hernia repairs. This technique is more reliable, solely performed by surgeons, and is supposed to replace the ultrasound-guided method. The latter is time-consuming, need ultrasound skills and is usually done by anaesthetists. Previous reports have shown advantage for the ultrasound-guided TAP block in controlling postoperative pain for several types of surgery. Our previous study for use of laparoscopically delivered TAP block in Laparoscopic Cholecystectomy has shown significant advantage in pain relief.

Among these, four trials have examined the beneficial effect of TAP block for inguinal hernia repair. Two studies controlled against placebo or no block groups, one compared TAP block with periportal infiltration, while another study compared single injection TAP block with continuous TAP block. Three studies used ultrasound to deliver the block. The Fourth study used semi-blind TAP blocks. One of the studies included open inguinal hernia repair as well.

The current trial is supposed to be the first one to evaluate the new method and comparing it with the current practice. In addition, the investigators will be using multi-modal analgesia.

Methodology:

Settings:

The study will be conducted in the Department of General surgery at Mayo University Hospital, Ireland.

Study design:

The current study is a prospective, randomized, Double-blinded parallel trial.

Study population:

Eighty six consecutive patients undergoing laparoscopic inguinal hernia repair (TEP) will be included in the study, 43 patients is each arm. One group will have surgically-assisted TAP block with bupivacaine and the others will have peri-portal local anesthetic infiltration. The patients will be randomized into two groups using "random number table" technique. The postoperative pain scoring will be recorded by two observers using numerical analog scale (NAS), but neither the patients nor the observers will be informed about the type of analgesia used.

Informed consent will be sought from all patients, and ethical approval will be sought from the institutional review board. The study will meet the standards outlined in the Declaration of Helsinki and Good practices. The trial will be registered at www.clinicaltrials.gov.

Sample size calculation:

SD of pain score = 1.83 (previous report by Mun Gyu Kim et al). Power = 90%. α = 0.05. Sample size per group = 43.

Surgery:

The surgery will be performed by one general surgeon following standardized surgical approach under general anaesthesia, while the TAP block will be done by one of the two surgeons who are familiar with the technique. The intra-abdominal pressure will be set at the same level (15 mm Hg) for all patients.

Intervention:

Test group:

The TAP block will be performed at lumbar triangle of petit (Triangle bounded by latissmus dorsi posteriorly, external oblique anteriorly and base by iliac crest) using a blunt needle. Local anaesthetic is injected at midaxillary line after establishing the space of Bogros (space between peritoneum and transversalis fascia). All the procedure will be performed under direct visualization of the laparoscope. Digital pressure will applied to define the site of injection. The needle will be inserted at the site of injection till it is short of transversalis fascia and slight tenting is visible . Then the plunger will be withdrawn to exclude vascular placement and the injection will be employed. The site of injection will be inspected from within the space of Bogros. The presence of internal bulge is regarded as the definitive point of the procedure.

Control group:

Local periportal infiltration will be done at the three ports before the insertion of ports.

Dosing:

Fixed dose of Bupivacaine (Total: 30 ml of 0.25% for the Test group and 15 ml of 0.5% for control group) will be given to all patients.

Test group: Angle of Petit ---- 30 ml of 0.25%. Control group: Camera port ---- 7 ml of 0.5%. Other ports ---- 4 ml of 0.5% each.

.

Postoperative pain management:

Standardized analgesic regimen will be used in the postoperative period. All patients will receive paracetamol 1000 mg / 6 hourly, orally + Dexketoprofen 50 mg (at 8 hrs).

For rescue analgesia: Tapentadol 75 mg/ As required. Total opiods used in peri operative period will be recorded.

Double blinding:

The patient and the observer will not know the control or intervention group.

Study end-points:

Primary: Pain score at rest and while coughing using the Numerical analog scale (NAS) at 1, 3, 6 and 24 hr.

Secondary: Analgesics requirements ( Paracetamol, NSAID and opiods). Nausea and vomiting.

Statistical analysis:

Group comparison will be done using Student t-test (2-tailed), Pearson chi-square test, and Mann-Whitney test. Alpha will be set at 0.05, and the SSPS 17.0 will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive ASA grade I-II- III patients undergoing elective unilateral laparoscopic total extra peritoneal (TEP) Inguinal hernia repair
* Age 18 - 80 yrs, including those who are having recurrent inguinal hernia repair.

Exclusion Criteria:

* ASA grade IV, V
* Bilateral inguinal hernia repair
* BMI > 40 kg/m2
* Converted to open procedures.
* Conversion to Transabdominal preperitoneal (TAPP) repair
* Coagulopathy.
* Allergy to Bupivacaine.
* Diagnosis of "chronic pain syndrome".
* Known alcohol or substance abuse within the last 6 months.
* Daily Opioid intake.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | Within 24 hours post surgery
  Numerical Analogue score for pain will be recorded at 1, 3, 6 and 24 hours post surgery

SECONDARY OUTCOMES:
Total opioid usage | within 24 hours perioperative period
  amount of opioids used in perioperative period will be recorded.
Post operative nausea or vomiting | 24 hours post operative period
  instances of nausea or vomiting in the post operative period will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Asif Khan, MBBS, MRCSI, Principal Investigator — Mayo University Hospital
Locations (1):
- Mayo University Hospital, Castlebar, Mayo, Ireland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Elamin G, Waters PS, Hamid H, O'Keeffe HM, Waldron RM, Duggan M, Khan W, Barry MK, Khan IZ. Efficacy of a Laparoscopically Delivered Transversus Abdominis Plane Block Technique during Elective Laparoscopic Cholecystectomy: A Prospective, Double-Blind Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):335-44. doi: 10.1016/j.jamcollsurg.2015.03.030. Epub 2015 Mar 27. PMID 25899736
- [Result] Chetwood A, Agrawal S, Hrouda D, Doyle P. Laparoscopic assisted transversus abdominis plane block: a novel insertion technique during laparoscopic nephrectomy. Anaesthesia. 2011 Apr;66(4):317-8. doi: 10.1111/j.1365-2044.2011.06664.x. No abstract available. PMID 21401554
- [Result] Kim MG, Kim SI, Ok SY, Kim SH, Lee SJ, Park SY, Yoo JH, Cho A, Hur KY, Kim MJ. Is transverse abdominis plane block effective following local anesthetic infiltration in laparoscopic totally extraperitoneal hernia repair? Korean J Anesthesiol. 2014 Dec;67(6):398-403. doi: 10.4097/kjae.2014.67.6.398. Epub 2014 Dec 29. PMID 25558340